CLINICAL TRIAL: NCT06483971
Title: Comparison of Oral Isotretinoin Versus Ancomparison of Oral Isotretinoin Versus Antibiotics on Corneal Thickness in Patients With Acne Vulgaris
Brief Title: Comparison of Oral Isotretinoin vs Ancomparison of Oral Isotretinoin vs Antibiotics on Corneal Thickness With AV
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MSRSW/Batch-Fall22/731
Record Dates: First submitted 2024-06-26; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Cornea
MeSH Terms: conditions — Corneal Diseases | interventions — Anti-Bacterial Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral Isotretinoin (Other)
  Interventions: Diagnostic Test: Oral Isotretinoin
- Antibiotics (Experimental)
  Interventions: Combination Product: Antibiotics

INTERVENTIONS:
Diagnostic Test: Oral Isotretinoin — 20 mg/kg/day that affects sebaceous glands and is used to treat severe acne Frequency: Once daily
  Arms: Oral Isotretinoin
Combination Product: Antibiotics — 250 mg on laternate day/3 months Frequency: Once or twice daily
  Arms: Antibiotics

SUMMARY:
Comparison of Oral Isotretinoin versus comparison of Oral Isotretinoin versus Antibiotics on Corneal Thickness in Patients with Acne Vulgaris

DETAILED DESCRIPTION:
Acne is the most common skin disease requiring attention of health practitioners. It is a self-limiting disease of the pilosebaceous unit, which can lead to devastating and frustrating scars and pigmentary alterations.

ELIGIBILITY:
Inclusion Criteria:

* Patients of either gender shall be enrolled for this study.
* Acne vulgaris patients taking oral isotretinoin and oral antibiotics shall be included.

Exclusion Criteria:

* Patients with any ocular pathology shall be excluded.
* Patients with any systemic pathology other than acne vulgaris shall be excluded.
* Patients with history of contact lens wear, previous refractive surgery or injury shall be excluded.

Ages: 20 Years to 43 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
Optical Coherence Tomography (OCT) | 12 Months
  Standardized OCT imaging protocols to ensure consistency and accuracy across all measurements.
Snellen Chart | 12 months
  Visual acuity measured at 3-month and 6-month intervals. Units: Snellen fraction (e.g., 20/20, 20/40)

CONTACTS AND LOCATIONS:
Locations (1):
- Shalamar Hospital Mughalpura, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No